CLINICAL TRIAL: NCT03058861
Title: Mitigating ACEs in Pediatric Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Seth Scholer, Associate Professor of Pediatrics, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB#161987
Record Dates: First submitted 2017-01-26; First posted 2017-02-23 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2024-02

CONDITIONS: Violence; Parenting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Discipline education - Play Nicely program (Experimental): Parents in the intervention group will receive 1) a copy of the Play Nicely Healthy Discipline Handbook (see www.playnicely.org), 2) information about how to view the Play Nicely multimedia program online and 3) the TN ACEs Handout.
  Interventions: Behavioral: Play Nicely Program
- Control Group (No Intervention): Routine primary care will be provided.

INTERVENTIONS:
Behavioral: Play Nicely Program — Play Nicely multimedia program and handbook that provides education about healthy discipline strategies.
  Arms: Discipline education - Play Nicely program

SUMMARY:
The project is designed to assess Adverse Childhood Experiences (ACEs) and test a parenting intervention in pediatric primary care.

DETAILED DESCRIPTION:
The goal of the project is to affect policy and practice related to Adverse Childhood Experiences (ACEs) screening and intervention in pediatric primary care. First, the investigators will develop and test a new ACEs screening tool that is brief, has a pediatric perspective, builds on parents' strengths, and measures parenting-related ACEs that can be treated. The new ACEs screening tool will measure parenting-related ACEs (e.g. corporal punishment, threatening, humiliation) and family stressors (e.g. divorce, incarceration, mental illness). A research assistant will invite approximately 1000 parents to complete the survey in the Vanderbilt Pediatric Primary Care Clinic. Measures will include child behavior problems that the investigators hypothesize will be associated with elevated parenting scores. The second part of the project will be to recruit English and Spanish-speaking parents for a randomized controlled trial (RCT) to determine if educational interventions can help educate parents about ACEs and decrease parenting-related ACE scores two months post-intervention. In the RCT, the investigators will recruit 300 to 400 parents to participate in the study. Parents in the intervention group will receive 1) a copy of the Play Nicely Healthy Discipline Handbook, 2) information about how to view the Play Nicely multimedia program online and 3) the TN ACEs Handout. Parents in the Control Group will receive routine primary care. Follow up data will be obtained 2 months after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Parents of 2-10 year old children presenting for a well visit.

Exclusion Criteria:

* Parents do not speak English, Spanish, or Arabic.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 576 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2018-01-03 (Actual); Study Completion 2018-01-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline Parenting Survey at 2 months | Baseline and 2 months
  Parenting Survey: 12 item scale that assesses parenting behaviors.

SECONDARY OUTCOMES:
Change from baseline Attitudes Toward Spanking scale at 2 months | Baseline and 2 months
  Attitudes Toward Spanking scale

CONTACTS AND LOCATIONS:
Overall Officials: Seth Scholer, MD,MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt Pediatric Primary Care Clinic, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sausen KA, Randolph JW, Casciato AN, Dietrich MS, Scholer SJ. The Development, Preliminary Validation, and Clinical Application of the Quick Parenting Assessment. Prev Sci. 2022 Feb;23(2):306-320. doi: 10.1007/s11121-021-01320-w. Epub 2021 Nov 15. PMID 34780005